CLINICAL TRIAL: NCT01308762
Title: An Intra-patient Placebo-controlled, Phase I Clinical Study, to Evaluate the Safety and Tolerability of Intradermal IMM-101 (Heat-killed Mycobacterium Obuense) in Adult Melanoma Cancer Patients
Brief Title: A Clinical Study, to Evaluate the Safety and Tolerability of Intradermal IMM-101 in Adult Melanoma Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immodulon Therapeutics Ltd (Industry)
Collaborators: HCA International Limited (Other); Theradex (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: IMM-101-001; 2009-012447-42 (EudraCT Number)
Record Dates: First submitted 2011-02-16; First posted 2011-03-04 (Estimated); Results first posted 2012-12-06 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-09

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — IMM-101

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMM-101 (Experimental): Patients received an intradermal injection of a single dose level of IMM 101 on three subsequent occasions. Doses of IMM 101 were administered over a 4 week period on days 0, 14 and 28. Doses used were:
  'Heat killed whole cell M. obuense (IMM-101) 0.1 mg', 'Heat killed whole cell M. obuense (IMM-101) 0.5 mg', or 'Heat killed whole cell M. obuense (IMM-101) 1.0 mg'
  Interventions: Biological: Heat killed whole cell M. obuense (IMM-101) 0.1 mg; Biological: Heat-killed whole cell M.obuense (IMM-101) 0.5 mg; Biological: Heat killed whole cell M.obuense (IMM-101) 1.0 mg

INTERVENTIONS:
Biological: Heat killed whole cell M. obuense (IMM-101) 0.1 mg — Each patient will receive an intradermal placebo injection of borate buffered saline solution (day -3) to provide an intra patient placebo control. Patients who were willing and able to proceed with the study will receive an intradermal injection of a single dose level of IMM 101 on three subsequent occasions. Doses of IMM 101 were administered over a 4 week period on days 0, 14 and 28.
  Dose levels to be administered are 0.1 mg, 0.5 mg and 1.0 mg.
  Other Names: IMM-101; Mycobaterium obuense
Biological: Heat-killed whole cell M.obuense (IMM-101) 0.5 mg — Each patient will receive an intradermal placebo injection of borate buffered saline solution (day -3) to provide an intra patient placebo control. Patients who were willing and able to proceed with the study will receive an intradermal injection of a single dose level of IMM 101 on three subsequent occasions. Doses of IMM 101 were administered over a 4 week period on days 0, 14 and 28.
  Other Names: IMM-101; Mycobaterium obuense
Biological: Heat killed whole cell M.obuense (IMM-101) 1.0 mg — Each patient will receive an intradermal placebo injection of borate buffered saline solution (day -3) to provide an intra patient placebo control. Patients who were willing and able to proceed with the study will receive an intradermal injection of a single dose level of IMM 101 on three subsequent occasions. Doses of IMM 101 were administered over a 4 week period on days 0, 14 and 28.
  Other Names: IMM-101; Mycobaterium obuense

SUMMARY:
To evaluate the safety and tolerability of intradermal injections of IMM-101 (Heat-killed Mycobacterium obuense) in melanoma cancer patients.

DETAILED DESCRIPTION:
The proposed study is a first-in-man, placebo-controlled, dose escalation trial to evaluate the safety and tolerability of three different doses of IMM-101 administered intradermally to melanoma patients. Additionally, the study aims to characterize local responses to this vaccine in order to delineate unexpected / unacceptable local reactions from those indicative of appropriate immunological response in this patient group.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of disease free stage III or stage IV melanoma (with or without metastases) or stable disease (if with metastases) and receiving no other treatment
* willing to use effective contraception for the duration of the study
* able to comply with the requirement to complete a diary card

Exclusion Criteria:

* Pregnant or lactating females
* Major surgery within the 14 days preceding the screening visit
* Suspicion of a previous infection with mycobacteria including previous tuberculosis (TB) prophylaxis
* Treatment with another investigational medicinal product within the last 30 days prior to the screening visit
* Previous treatment with M. vaccae
* Exposure to Bacille Calmette Guérin vaccine (BCG) within the last 12 months
* Concurrent uses of drugs likely to reduce inflammation at the local injection site or dampen/modulate the immune system
* Depot injection of corticosteroids within 6 weeks of the screening visit or chronic systemic corticosteroids in the 2 weeks prior to the screening visit
* Ongoing treatment with radiotherapy, cytotoxic chemotherapy or chemotherapy in the last 30 days prior to the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Stebbings, Professor, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- HCA Clinical Trials Unit, 79 Harley Street,, London, United Kingdom

REFERENCES:
- [Derived] Stebbing J, Dalgleish A, Gifford-Moore A, Martin A, Gleeson C, Wilson G, Brunet LR, Grange J, Mudan S. An intra-patient placebo-controlled phase I trial to evaluate the safety and tolerability of intradermal IMM-101 in melanoma. Ann Oncol. 2012 May;23(5):1314-1319. doi: 10.1093/annonc/mdr363. Epub 2011 Sep 19. PMID 21930686

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 24 patients with melanoma entered the screening phase of this study between 10 March 2010 and 27 July 2010.
Pre-assignment Details: Five patients were found to be ineligible and failed screening. These patients were withdrawn before receiving study medication.
Groups:
- IMM-101 0.1 mg: Patients received an intradermal injection of IMM-101 0.1 mg on three occasions. Doses were administered over a four week period on days 0, 14 and 28.
- IMM-101 0.5 mg: Patients received an intradermal injection of IMM-101 0.5 mg on three occasions. Doses were administered over a four week period on days 0, 14 and 28.
- IMM-101 1.0 mg: Patients received an intradermal injection of IMM-101 1.0 mg on three occasions. Doses were administered over a four week period on days 0, 14 and 28.
Period: Overall Study
Arm/Group | IMM-101 0.1 mg | IMM-101 0.5 mg | IMM-101 1.0 mg
Started | 6 | 7 | 6
Completed | 6 | 6 (One patient was withdrawn as they were retrospecively found to have been ineligible at study entry) | 6
Not Completed | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: IMM-101 0.1 mg
- Group 2: IMM-101 0.5 mg
- Group 3: IMM-101 1.0 mg
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 6 | 7 | 6 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 3 | 11
  >=65 years | 1 | 4 | 3 | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 47.3 (17.3) | 56.1 (20.2) | 56.3 (18.8) | 53.4 (18.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 8
  Male | 4 | 4 | 3 | 11
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 7 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Safety and tolerability were measured with respect to:
  1. Safety measurements
  2. Local tolerability at the site of intradermal injection
  3. Incidence of adverse events.
Time Frame: 56 days
Population: All analyses were based on the safety population, which comprised of all patients who received at least one dose of IMP. Safety measurements and nature and incidence of adverse events were reported for the Safety population
Measure: Number; unit: Participants
Groups:
- IMM-101 0.1 mg; IMM-101 0.5 mg; IMM-101 1.0 mg: IMM-101 was administered on 3 separate occasions to the same individual over a 4 week period (Day 1, 14 and 28).
Arm/Group | IMM-101 0.1 mg | IMM-101 0.5 mg | IMM-101 1.0 mg
Number analyzed (Participants) | 6 | 7 | 6
Participants | 6 | 7 | 6

2. Secondary Outcome: Administration Site Reactions
Description: Local skin reactions are viewed as a normal and predicted reaction to exposure to a preparation of mycobacterial antigens. All patients experienced administration site reactions and all reactions were examined and characterised. However only those reported as adverse events are presented here.
Time Frame: Day -3 to Day 56
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 6 | 7 | 6
Participants | 1 | 3 | 5

ADVERSE EVENTS:
Time Frame: Adverse event data were collected on the followings days: -3, 0, 3, 14, 17, 28, 31, 42, 56
Description: In accordance with the EU Clinical Trials Directive the investigator reported any directly observed AEs and any AEs reported spontaneously by the patient. In addition, each patient was questioned about AEs at each visit before administration of study medication.
Arm/Group | Group 1 | Group 2 | Group 3
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/7 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 7/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=6) | Group 2 (N=7) | Group 3 (N=6)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Patient experienced progressive shortness of breath and was hospitalised for supportive care whilst undergoing investigations. The cause was collapse of the left lower lobe of the lung with a metastatic mass - consistent with progressive disease.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=6) | Group 2 (N=7) | Group 3 (N=6)
Altered ECG (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Common cold (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Enlarged Lymph node (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Eye proptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Flu-like symptoms (General disorders) | 2 (2) | 2 (3) | 2 (3)
Generalised or joint ache /pain (General disorders) | 3 (3) | 4 (11) | 5 (11)
Hard red swelling on cheek (General disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 4 (8)
Herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hypotension (General disorders) | 0 (0) | 2 (2) | 0 (0)
Increased LDH (Investigations) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (5) | 3 (5) | 5 (19)
Mild ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
New Lump (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
New lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Red eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Redness on face (General disorders) | 1 (1) | 0 (0) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Skin erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Temperature (General disorders) | 0 (0) | 2 (3) | 2 (3)
Tiredness (General disorders) | 1 (1) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Warts (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less